CLINICAL TRIAL: NCT04864119
Title: DEFINing the PrEvalence and Characteristics of Coronary Artery Disease Among Patients With TYPE 2 Myocardial Infarction Using CT-FFR
Acronym: DEFINE TYPE2MI
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: HeartFlow, Inc. (Industry)
Responsible Party: Principal Investigator, James L. Januzzi, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2021P000435
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives of this study include:

* determine the prevalence of coronary artery disease among patients with type 2 myocardial infarction
* determine the prevalence of hemodynamically significant stenosis among patients with type 2 myocardial infarction

The investigators hypothesize that patients with type 2 myocardial infarction will have a high burden of coronary artery plaque and a high prevalence of obstructive coronary artery disease with hemodynamic significance.

DETAILED DESCRIPTION:
RECRUITMENT

Patients in the Emergency Department or admitted to Massachusetts General Hospital with an elevated high-sensitivity cardiac troponin will be identified daily by the Clinical Core Laboratory at Massachusetts General Hospital. The study investigators will then review the electronic medical record for each of these patients to determine if the cause of the patients' elevated high-sensitivity troponin is a type 2 myocardial infarction. If so, their record will be reviewed to determine if they meet the inclusion criteria for enrollment and to ensure no exclusion criteria are present. Patients with a type 2 MI who are eligible for enrollment, will then be approached during their hospital stay to discuss the study and their interest in consenting and enrolling in our study. Prior to approaching the patient, the responding clinician treating the patient will be contacted to obtain the primary team's approval before approaching the patient. In addition to confirming that the patient is an acceptable candidate for the research, a clinician from the primary team must introduce the study to the patient and obtain the patient's permission prior to being contacted by our study staff. 50 patients will be enrolled.

STUDY PROCEDURES

1. Study visits and parameters to be measured (e.g. laboratory tests, x-rays, and other testing) Patients who enroll in the study will undergo a CT coronary angiogram during their index admission. In addition, patients will have the option of providing a blood sample for future research. These biorepository samples may be used in the future for biomarker analysis to examine associations between serum biomarkers of cardiac injury, inflammation, and atherosclerosis, and coronary plaque presence/ severity and for predicting future cardiovascular events up to 1-year. Genetic testing will not be performed on these samples. There will be no required follow-up visits following their index admission.
2. Drugs to be used (dose, method, schedule of administration, dose modifications, toxicities).

   Patients will receive nitroglycerin prior to their CT coronary angiogram in the form of a transdermal patch (0.8 mg/h [2 x 0.4 mg/h]; Nitro-Dur, Merck & Co. Inc., White-House Station, New Jersey). Nitroglycerin will be administered at least 45 minutes before electrocardiography-gated coronary CTA.

   Iohexol (OMNIPAQUE-350) 350 mg iodine/ml solution 150ml will be used as an iodinated contrast agent for the scan as per standard protocol at our institution.
3. Devices to be used Patients will undergo a CT coronary angiogram. Once the images are obtained, they will be sent to HeartFlow Inc for fractional flow analysis using their FDA-approved CT-FFR software.
4. Procedures/surgical interventions, etc. As this is a prospective observational study, no procedures or interventions will be made. Any significant findings from the CT scan will be relayed to the patient and the medical team.
5. Data to be collected and when it will be collected

For patients who enroll in this study, the following information will be collected during their index admission:

Demographic information Past Medical History Home cardiac medications Cause of type 2 myocardial infarction Laboratory information Cardiac testing Results of CT coronary angiogram including presence and severity of coronary artery disease, total coronary plaque volume, calcified plaque volume, non-calcified plaque volume, and LV mass Results of CT-FFR Results of invasive coronary angiogram (including intravascular ultrasound and optical coherence tomography) if performed In-hospital outcomes including mortality, acute kidney injury, recurrent MI, and stroke Discharge cardiac medications

Following discharge:

Using the electronic medical record, the following data will be collected via chart review:

1-year outcomes including all-cause hospital readmission, recurrent MI, heart failure hospitalization, stroke, and mortality.

Source of subjects and recruitment methods To screen for patients with type 2 MI the investigators will first identify patients at Massachusetts General Hospital with an elevated high-sensitivity cardiac troponin on a daily basis through the MGH Central Laboratory. For patients with elevated troponin, the investigators will review their medical records to determine if the cause of their troponin elevation is a type 2 MI. For patients with type 2 MI, their medical record will be reviewed to ensure there are eligible for enrollment based on our inclusion and exclusion criteria.

BIOSTATISCAL ANALYSIS

a. Specific data variables being collected for the study During the index hospitalization Demographic information Past Medical History Home cardiac medications Cause of type 2 myocardial infarction Laboratory information Cardiac testing Results of CT coronary angiogram including presence and severity of coronary artery disease, total coronary plaque volume, calcified plaque volume, non-calcified plaque volume, and LV mass Results of CT-FFR Results of invasive coronary angiogram (including intravascular ultrasound and optical coherence tomography) if performed In-hospital outcomes including mortality, acute kidney injury, recurrent MI, and stroke Discharge cardiac medications

Following discharge:

Using the electronic medical record, the following data will be collected via chart review:

1-year outcomes including all-cause hospital readmission, recurrent MI, heart failure hospitalization, stroke, and mortality.

DATA & SAFETY MONITORING The principal investigator will review any adverse events that occur during the CT coronary angiogram. This will involve reviewing the patient's medical record for any serious or life-threatening allergic reactions, kidney injury from contrast material necessitating initiation of dialysis, and serious adverse reactions to nitroglycerin. This review will occur monthly.

Unanticipated problems involving risks to subjects or others including adverse events will be reported to the study sponsor and the Partners Human Research Committee (IRB) by the Principal Investigator within 5 working days (7 calendar days) in accordance with Partners Human Research Committee unanticipated problems including adverse events reporting guidelines.

Drs. McCarthy and Januzzi will be responsible for monitoring the accuracy and completeness of case report form entries into REDCap and the informed consent forms.

PRIVACY & CONFIDENTIALITY

Study data will be collected and stored on Partners REDCap (Research Electronic Data Capture), a secure, electronic SSL-encrypted, web-based application. Only study investigators will have access to the data.

Blood samples obtained will be stored on-site at Massachusetts General Hospital in a secure location.

Deidentified data collected by study investigators may be shared with the study Sponsor. This may include patient demographic data, medical history, cardiac test results, and patient outcomes. No identifiable data or sensitive information will be shared with the Sponsor. As this is a single-center study, no data will be shared with other collaborators outside of Partners. No specimens or data will be stored at collaborating sites outside of partners.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent
* Patients aged greater than18 years diagnosed with type 2 MI, defined based on the 4th Universal Definition of Myocardial Infarction (1), during their index hospitalization
* Type 2 MI will be defined as detection of a rise and/or fall of troponin levels with at least one value above the 99th percentile and evidence of an imbalance between myocardial oxygen supply and demand, requiring at least one of the following:

  * Symptoms of acute myocardial ischemia;
  * New ischemic ECG changes;
  * Development of pathological Q waves;
  * Imaging evidence of new loss of viable myocardium, or new regional wall motion abnormality in a pattern consistent with an ischemic etiology
* Patients with medical precipitants of their type 2 MI or post-operative type 2 MI. A minimum of 10 patients with post-operative type 2 MI will be included to ensure a diverse clinical patient population is enrolled.

Exclusion Criteria:

* Other types of MI
* Hemodynamic instability
* eGFR <30 ml/min/1.73m2
* Pregnant or breast-feeding women
* Contrast allergy
* Pre-operative history of MI, coronary angiography or coronary revascularization for patients with post-operative type 2 MI
* Severe arrhythmias precluding optimal CT image acquisition
* Prior coronary artery bypass grafting
* Known prior left main coronary artery PCI
* Known PCI of the left coronary system combined with >30% stenosis in the left main artery
* Known prior PCI to 2 or more major coronary vessels (i.e. left anterior descending artery, left circumflex artery, right coronary artery)
* Allergy or contraindication to nitroglycerin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a single-center prospective observational study that will enroll 50 adult patients who are admitted with a type 2 myocardial infarction at Massachusetts General Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-04-11 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of obstructive coronary artery disease | 1 year
  (defined as a stenosis of greater or equal to 70% in any epicardial vessel except left main coronary artery where greater or equal to 50% will be considered obstructive)
Prevalence of hemodynamically significant stenosis | 1 year
  as determined by FFR <0.8

SECONDARY OUTCOMES:
Prevalence of non-calcified coronary plaque | 1 year
Prevalence of high-risk plaque features | 1 year
Prevalence of any coronary plaque | 1 year
Prevalence of calcified coronary plaque | 1 year
Number of obstructive stenosis in coronary arteries | 1 year
Change in prescription rates for antiplatelet agents, lipid lowering therapy, beta blockers, and ACEi/ARB after CT coronary angiogram | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: James L Januzzi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
As this study will inform how often patients with this form of heart attack have coronary artery disease, this study will help inform us if we should be screening for coronary artery disease more frequently in patients with this form of heart attack.

REFERENCES:
- [Derived] Lin C, McCarthy CP, Mohebi R, Liu Y, Blankstein R, Murphy SP, Miksenas H, Rogers C, Amponsah DK, Rambarat PK, Raghavan A, Levin A, Ghoshhajra B, Wasfy JH, Hedgire S, Januzzi JL Jr. Sex Differences in Coronary Artery Disease Characteristics Among Patients With Type 2 Myocardial Infarction. JACC Adv. 2023 Dec 22;3(2):100795. doi: 10.1016/j.jacadv.2023.100795. eCollection 2024 Feb. PMID 38939381
- [Derived] McCarthy CP, Murphy SP, Amponsah DK, Rambarat PK, Lin C, Liu Y, Mohebi R, Levin A, Raghavan A, Miksenas H, Rogers C, Wasfy JH, Blankstein R, Ghoshhajra B, Hedgire S, Januzzi JL Jr. Coronary Computed Tomographic Angiography With Fractional Flow Reserve in Patients With Type 2 Myocardial Infarction. J Am Coll Cardiol. 2023 Oct 24;82(17):1676-1687. doi: 10.1016/j.jacc.2023.08.020. Epub 2023 Sep 29. PMID 37777947